CLINICAL TRIAL: NCT06716606
Title: An Open Label Study to Investigate the Long-term Safety and Efficacy of Belimumab in Adults With Interstitial Lung Disease (ILD) Associated With Systemic Sclerosis (SSc) and Other Connective Tissue Diseases (CTD)
Brief Title: A Study to Investigate the Long-term Safety and Efficacy of Belimumab in Adults With Interstitial Lung Disease (ILD) Associated With Systemic Sclerosis (SSc) and Other Connective Tissue Diseases (CTD) (BLISSconneCTD-OLE)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 219855; 2023-509370-39 (Other: EU CT Number)
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Connective Tissue Diseases
Keywords: Belimumab; Long-term; Open label extension; Interstitial lung disease; Diffuse cutaneous systemic sclerosis; Connective tissue disease
MeSH Terms: conditions — Connective Tissue Diseases; Lung Diseases, Interstitial; Scleroderma, Diffuse | interventions — belimumab

STUDY DESIGN:
Masking Description: This will be an Open Label Extension study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving Belimumab (Experimental): Participants will receive belimumab.
  Interventions: Drug: Belimumab

INTERVENTIONS:
Drug: Belimumab — Belimumab will be administered.

SUMMARY:
This is an open label extension (OLE) study of an ongoing randomized controlled parent clinical studies 218224 (NCT05878717) and 221672 (NCT06572384) which aim to assess the efficacy and safety of belimumab on reducing the decline in lung function in participants with interstitial lung disease associated with diffuse cutaneous systemic sclerosis (dcSSc-ILD) and interstitial lung disease associated with other connective tissue diseases (CTD-ILD), respectively. The OLE study will describe how well tolerated belimumab will be long term, and whether it might continue to slow progression of lung function decline, slow overall disease progression and improve quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Participants with SSc-ILD or other CTD-ILDs that have completed either study 218224 or 221672 through to and including the Week 52 visit and are not considered treatment failure, defined as meeting either of the following criteria:

  * Discontinuation of study medication during study 218224 or 221672 for any reason.
* Participants with SSc should have an area of uninvolved or mildly thickened skin that, in the opinion of the investigator, would allow subcutaneous (SC) injection at the abdomen or the front, middle region of the thigh.
* Participant is capable and willing to self-administer the study medication or has a caregiver/healthcare professional who is capable and willing to administer the study medication throughout the study.
* Female participants: A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

Is a woman of non-childbearing potential (WONCBP) or is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective, with a failure rate of less than (<)1 percentage (%), during the study treatment period and for at least 4 months after the last dose of study intervention. The investigator should evaluate potential for contraceptive method failure (e.g., non-compliance, recently initiated) in relationship to the first dose of study intervention.

1. A WOCBP must have a negative highly sensitive pregnancy test (urine or serum, as required by local regulations) within 24 hours before the first dose of study intervention.
2. If a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
3. Additional requirements for pregnancy testing during and after study intervention are located.
4. The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.

   * Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

* Participants of study 218224 or study 221672 who have discontinued study treatment, prior to Week 52.
* Participants who have developed clinical evidence of significant, unstable or uncontrolled, acute or chronic diseases not due to SSc or other CTD (i.e, cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases), or experienced an AE in study 218224 or study 221672 that could, in the opinion of the principal investigator, put the participant at undue risk.
* Participants who have developed any other medical diseases (eg, cardiopulmonary), laboratory abnormalities, or conditions (eg, poor venous access) that, in the opinion of the investigator could significantly alter the absorption, metabolism, or elimination of drugs; constitutes a risk when taking the study intervention; interferes with the interpretation of data; or it is not safe for the participant to continue on the study.
* Participants who have been exposed to ionizing radiation in excess of 10 millisievert (mSv) above background over the previous 3 year period as a result of occupational exposure or previous participation in research studies.
* QT Interval Corrected (QTc) greater than (>) 480 millisecond (msec) at Week 52 of parent study 218224 or study 221672.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-12-27 (Estimated); Study Completion 2029-12-27 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse events (AEs), Adverse Event of Special Interest events (AESIs), and Serious Adverse Event (SAEs) | Up to approximately 5 years

SECONDARY OUTCOMES:
Change from Baseline in Forced Vital Capacity (FVC) | Baseline (Day 1 of OLE study) and at Weeks 12, 26 and 52

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- GSK Investigational Site, Philadelphia, Pennsylvania, United States
- Argentina (2):
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
- China (2):
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Zhuzhou
- GSK Investigational Site, Larissa, Greece
- Japan (2):
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Yongsan-Ku Seoul, South Korea
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/